CLINICAL TRIAL: NCT03796091
Title: Efficacy Trial of a Dissonance Based Eating Disorder Program
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cornell College (Other)
Collaborators: National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Dr. Melinda Green, Principal Investigator, Cornell College
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 1516-105-GRE; R15MH113044 (NIH)
Record Dates: First submitted 2018-12-31; First posted 2019-01-08 (Actual); Results first posted 2022-12-09 (Actual); Last update posted 2022-12-09 (Actual); Status verified 2022-11

CONDITIONS: Eating Disorder
MeSH Terms: conditions — Feeding and Eating Disorders

STUDY DESIGN:
Intervention Model Description: Randomized, controlled clinical trial with 3 treatment interventions
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Educational Brochure (Active Comparator): Participants will read an educational brochure from the National Eating Disorder Association and will receive referral resources.
  Interventions: Behavioral: Educational Brochure
- Body Project Traditional (Active Comparator): Participants will complete group therapy for 1-hour per week for 4 weeks consisting of the Body Project group therapy program (Stice & Shaw, 2001).
  Interventions: Behavioral: Body Project Traditional
- Body Project Expanded (Active Comparator): Participants will complete group therapy for 1-hour per week for 4 weeks consisting of the Body Project Expanded group therapy program (Green et al., 2017).
  Interventions: Behavioral: Body Project Expanded

INTERVENTIONS:
Behavioral: Educational Brochure — Participants will read an educational brochure from the National Eating Disorders Association and will receive treatment referral resources.
  Arms: Educational Brochure
Behavioral: Body Project Traditional — Participants will complete a 1-hour per week group therapy program for 4 weeks consisting of the Body Project Traditional group therapy program (see Stice & Shaw, 2001).
  Arms: Body Project Traditional
Behavioral: Body Project Expanded — Participants will complete a 1-hour per week group therapy program for 4 weeks consisting of the Body Project Expanded group therapy program (see Green et al., 2017).
  Arms: Body Project Expanded

SUMMARY:
The purpose of this clinical trial is to investigate whether symptoms of disordered eating change among participants who complete an intervention. Participants will be randomly assigned to one of three intervention conditions and will undergo assessments of symptoms before, after, and 2 months after each intervention. Investigators are evaluating which interventions are most effective in reducing eating disorder symptoms and disorder-related psychological and cardiac risk factors.

DETAILED DESCRIPTION:
Assessment Sessions (Preintervention, Postintervention, 2-month follow-up): Participants in all conditions will participate in a series of 3 assessment sessions. Prior to each session, participants will complete online questions assessing eating disorder symptoms and associated psychological risk factors. This process will take approximately 40 minutes. Next participants will report to the laboratory at their scheduled appointment time to have their cardiac function assessed via blood pressure measurements and electrocardiography (EKG or ECG). Participants' height and weight will also be recorded.

Prior to each assessment session, participants should:

* Complete the online survey (if not completed prior to each laboratory appointment this will need to be completed at the lab appointment)
* Fast (not consume any food or beverages other than water) for at least 3 hours.
* Refrain from using nicotine for at least 3 hours.
* Refrain from vigorous physical exercise for at least 24 hours.
* Not show any symptoms of acute physical illness for 48 hours. It is important for participants to follow these directions so researchers can gather the most accurate data. If participants forget to follow these guidelines, or if an illness occurs, participants should contact their experimenter to reschedule.

On the day of an assessment session, participants will drive to the assessment location. Participants will receive directions via e-mail prior to each session. During the assessment session, participants will lie down on a laboratory cot for 10 minutes while preparation for electrocardiography (EKG or ECG) occurs. Electrodes will be applied to the chest and torso and lead wires will be attached to the electrodes. Participants' blood pressure will be assessed several times throughout this interval. Next, the experimenter will collect a 5 minute and 30 second recording of participants' cardiovascular data via electrocardiography (ECG or EKG). This data will later be analyzed to examine cardiac function.Next experimenters will assess participants' height and weight.

After each assessment session, participants' eating disorder symptoms, psychological risk factors, and cardiac indices will be evaluated by the research team. If the team determines that symptoms or cardiac indices are atypical and indicate a further need for evaluation, the participant will be contacted via both e-mail and phone to be informed results are atypical and the participant will be referred for further evaluation by a medical provider. If the participant is a minor, this information will be provided both to the participant and to the participant's parent and/or the participant's legal guardian. If participants' symptoms or risk factors worsen significantly over the duration of the trial, participants will also be contacted and provided with referral recommendations.

All participants will receive a comprehensive symptom report at the end of the trial. Referral resources will be provided again at that time if significant eating disorder symptoms remain.

Treatment Conditions: Participants will be randomly assigned to 1 of 3 treatment conditions.

Brochure Treatment Condition: Participants randomly assigned to the educational brochure will receive two educational brochures which discuss eating disorder symptoms. The brochures will also include treatment referral information and recommended resources for persons struggling with disordered eating. The brochure will take approximately 10 minutes to read; follow-up with treatment or self-help referral resources is completely voluntary.

Group Therapy Treatment Conditions: Participants randomly assigned to one of the two group treatment intervention conditions will complete a 4-week group treatment program with 3-8 other women and 2 trained treatment co-facilitators. For approximately 1 hour each week, participants will meet in this group to complete a series of readings, written activities, and verbal activities designed to reduce disordered eating. During the 4 intervention sessions, participants will be asked to analyze the weight and appearance-related messages received from the media, peers, family, romantic partners, and other sources. Participants will also be asked to record, analyze, and evaluate weight and appearance-related thoughts, emotions, and behaviors. Participants will engage in a variety of exercises designed to evaluate the meaning of thinness in our culture and its personal impact. These exercises are designed to combat the detrimental impact of messages which promote thinness.

Other risk factors will also be addressed, depending upon program. Participants may talk about the pressures women receive to focus on appearance. The relationship between these appearance-related pressures and eating disorder symptoms will be explored. Participants will explore the way they compare themselves to others and participate in a series of discussions and activities designed to decrease appearance-based comparisons with others.

After the 4-week program is complete, participants in both intervention conditions will continue to work on homework assignments related to the program for a period of 2-months until the final assessment session.

ELIGIBILITY:
Inclusion Criteria:

* Inclusion Criteria

  * Women
  * Age 15-34
  * Postmenarcheal
  * Premenopausal
  * Subclinical or Clinical Eating Disorder Symptoms

Exclusion Criteria:

* Exclusion Criteria

  * Must get physician clearance to participate if at medically high risk as defined in the protocol
  * Must not be pregnant
  * Must be able to read and speak English

Ages: 15 Years to 34 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 180 (Actual)
Dates: Start 2018-11-18 (Actual); Primary Completion 2021-04-15 (Actual); Study Completion 2021-04-15 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Melinda A Green, PhD, Principal Investigator — Green Counseling Services PLLC
Locations (1):
- Cornell College Eating Disorder Institute, Mount Vernon, Iowa, United States

IPD SHARING:
Plan to Share IPD: Yes
Data will be made available to other researchers upon request and subject to signed confidentiality agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: Upon request with 5 years of study completion.
Access Criteria: Must sign confidentiality agreement.

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Women aged 15-35 displaying subclinical and clinical eating disorder symptoms were recruited from 2 Midwestern cities and 5 surrounding suburban communities from November of 2018 to March of 2021. All participants were treated in accordance with federal guidelines (Title 45, Code of Regulations Part 46) for the treatment of human participants. The research was approved by an Institutional Review Board at the host institution.
Pre-assignment Details: All participants were screened to ensure inclusion criteria were met. Inclusion criteria specified female participants ages 15-34 (postmenarcheal and premenopausal) who were not pregnant. Participant selection was limited to this group to control for the effects of estrogen on cardiac function and in accordance with previous research which suggests dissonance-based programs are most effective when offered solely to females over the age of 15.
Period: Overall Study
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Started | 60 | 60 | 60
Completed | 40 | 38 | 45
Not Completed | 20 | 22 | 15

BASELINE CHARACTERISTICS:
Population: The numbers presented in the Baseline Analysis Population indicate the number of participants as a function of condition who completed the baseline assessment session. This differs from the number of participants in the Participant Flow Module because that module reflects the number of participants who completed the pre-trial screening and were enrolled in the trial. The discrepancy is explained by participants not attending the baseline assessment following study enrollment at screening.
Groups:
- Total: Total of all reporting groups
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded | Total
Number analyzed (Participants) | 49 | 51 | 50 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 22.48 (3.63) | 23.95 (5.73) | 21.73 (4.08) | 22.75 (4.65)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49 | 51 | 50 | 150
  Male | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 1 | 1 | 2
  Asian | 0 | 2 | 1 | 3
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 2 | 2 | 6 | 10
  White | 42 | 42 | 38 | 122
  More than one race | 4 | 3 | 1 | 8
  Unknown or Not Reported | 1 | 1 | 3 | 5
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 49 | 51 | 50 | 150
Rosenberg Self-Esteem Scale [Mean (Standard Deviation); unit: units on a scale] — The Rosenberg Self-Esteem Scale is designed to assess global feelings of self-worth. The RSE includes 10 items (e.g. "I feel that I'm a person of worth'') rated on a four-point scale (1 = strongly disagree, 4 = strongly agree). A total score represents the sum of individual item responses. Scores range from 10 to 40 and higher scores indicate higher levels of self-esteem.
  units on a scale | 22.71 (4.71) | 22.50 (4.81) | 22.62 (4.07) | 22.61 (4.53)
Eating Disorder Examination Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The 28-item Eating Disorder Examination Questionnaire global score was used to measure eating disorder symptomatology. Participants report symptomatology over the past 28 days on a 7-point Likert scale from 0 (no days) to 6 (everyday). The EDE-Q contains 4 subscales: Restraint, Weight Concern, Eating Concern, and Shape Concern. Subscale scores are calculated by finding the averages of the subscale items. A global score is also calculated by averaging the subscale scores. Scores range from 0 to 6; higher scores indicate higher levels of eating disorder pathology.
  units on a scale | 4.25 (0.8) | 3.93 (1.15) | 3.96 (1.02) | 4.04 (1.00)
Body Shape Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Body Shape Questionnaire (BSQ) was used to measure body dissatisfaction in the present trial. The BSQ is a 34-item scale. Items are measured on a 6-point Likert scale designed to assess the frequency of negative body-related thoughts (1= never, 6 = always). Individual items are summed to compute an overall score. Scores on this scale range from 34 to 204. Higher scores indicate higher frequency of negative body-related thoughts and higher levels of body dissatisfaction.
  units on a scale | 139.42 (23.92) | 134.37 (30.15) | 134.73 (28.32) | 136.17 (27.55)
Social Comparison Rating Scale [Mean (Standard Deviation); unit: units on a scale] — The Social Comparison Rating Scale (SCRS is an 11-item scale used to assess perception of social rank and social comparison tendencies in the present trial. The scale consists of a series of bipolar adjectives (e.g., inferior/superior) separated by the numbers 1 through 10. For each adjective pair, participants are asked to rank themselves in comparison to others. A score around 60 indicates a person, on average, sees themselves approximately equal to others. Higher scores indicate higher levels of favorable social comparison and higher perceived social rank.
  units on a scale | 45.59 (17.10) | 43.83 (13.18) | 43.00 (13.80) | 44.15 (14.75)
Self-Objectification Questionnaire [Mean (Standard Deviation); unit: units on a scale] — The Self-Objectification Questionnaire (SOQ) is a 10-item self-report inventory designed to assess the relative importance of body competence versus body appearance in sense of self. Participants rank appearance- versus competence-based attributes from 0 to 9 with higher scores representing higher importance. An overall trait self-objectification score is computed by summing competence and appearance ratings and subtracting the sum of competence ratings from the sum of appearance ratings. Resulting scores range from -25 to 25. Higher scores denote higher levels of trait self-objectification.
  units on a scale | 10.13 (9.75) | 7.71 (13.11) | 6.32 (12.46) | 8.07 (11.91)
Ideal Body Stereotype Scale Revised [Mean (Standard Deviation); unit: units on a scale] — The Ideal Body Stereotype Scale - Revised was used to assess the extent to which participants internalized the cultural feminine thin-ideal. The IBSS-R is a self-report inventory which asks participants to report their level of agreement with 6 statements which indicate what attractive women look like on a 5-point scale ranging from strongly disagree (1) to strongly agree (5). Responses are averaged to compute a total score. Scores ranges from 1 to 5; higher scores indicate higher levels of thin-ideal internalization.
  units on a scale | 3.81 (0.5) | 3.82 (.45) | 3.76 (0.5) | 3.79 (.48)
State Trait Anxiety Inventory Form Y [Mean (Standard Deviation); unit: units on a scale] — The State Trait Anxiety Inventory- Form Y (STAI) is a 20-item self-report measure used to assess level of trait anxiety in the present study. Each item consists of a statement which assesses feelings of anxiety or relaxation on a 4-point scale ranging from 1 (not at all) to 4 (very much so). Responses to individual items are summed to create an overall score. Scores range from 20 to 80. Higher scores indicate higher levels of anxiety.
  units on a scale | 58.87 (8.42) | 58.02 (7.84) | 58.70 (7.90) | 58.52 (7.84)
Positive and Negative Affect Scale - Positive Affect [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Affect Schedule is a 20-item self-report questionnaire that used to measure positive and negative affect. Items are rated on a 5-point scale ranging from 1 (very slightly) to 5 (extremely) which measures the extent to which the client has experienced that affect over the past week. The 10 positive and 10 negative items are summed separately to create a positive affect score and a negative affect score respectively. Each score ranges between 0 and 50 with higher scores indicating higher positive or negative affect.
  units on a scale | 26.35 (5.76) | 25.53 (7.10) | 25.24 (6.46) | 25.71 (6.45)
Mean R Wave Amplitude [Mean (Standard Deviation); unit: mV] — Mean R wave amplitude was determined via a 3-lead ECG and was measured in millivolts (mV). The ECG signal was acquired via PowerLab 16/35 psychophysiological data acquisition system with a sampling rate of 1000 Hz. Hardware setup included an ECG100C amplifier with a 35Hz LPN filter and a .5Hz HP filter. ECG data were analyzed via PowerLab LabChart 8 software. A total of 5 minutes and 30 seconds of ECG data were collected to allow for artifact trimming. Artifacts were flagged by experimenters during data collection.
  mV | 1.27 (.36) | 1.19 (.31) | 1.24 (.37) | 1.23 (.35)
QTc Prolongation [Mean (Standard Deviation); unit: msec] — QTc prolongation was measured in msec and was assessed via 3-lead ECG. The ECG signal was acquired via PowerLab 16/35 psychophysiological data acquisition system with a sampling rate of 1000 Hz. Hardware setup included an ECG100C amplifier with a 35Hz LPN filter and a .5Hz HP filter. ECG data were analyzed via PowerLab LabChart 8 software. For detection, typical QRS width was set at 80ms and R waves were at least 300ms apart. QTc was corrected with Bazett's formula.
  msec | .38 (.02) | .38 (.02) | .38 (.02) | .38 (.02)
Positive and Negative Affect Scale - Negative Affect [Mean (Standard Deviation); unit: units on a scale] — The Positive and Negative Affect Schedule is a 20-item self-report questionnaire that used to measure positive and negative affect. Items are rated on a 5-point scale ranging from 1 (very slightly) to 5 (extremely) which measures the extent to which the client has experienced that affect over the past week. The 10 positive and 10 negative items are summed separately to create a positive affect score and a negative affect score respectively. Each score ranges between 0 and 50 with higher scores indicating higher positive or negative affect.
  units on a scale | 30.15 (7.46) | 29.00 (6.88) | 29.64 (6.60) | 29.59 (6.97)
Vagal Cardiac Tone - High Frequency Spectral Power [Mean (Standard Deviation); unit: Normalized units: HF (watts/Hz)] — Vagal tone was assessed via heart rate variability (HRV) power spectral analysis of 3-lead ECG data and was reported in normalized units. The ECG signal was acquired via PowerLab 16/35 psychophysiological data acquisition system with a sampling rate of 1000 Hz. Hardware setup included an ECG100C amplifier with a 35Hz LPN filter and a .5Hz HP filter. ECG data were analyzed via PowerLab LabChart 8 software. Maximum frequency was set at 0.5 Hz with number of frequencies at 500. LF spectral power ranged from 0.04-0.15 Hz. HF spectral power ranged from 0.15-0.45 Hz.
  Normalized units: HF (watts/Hz) | 60.08 (19.56) | 57.26 (19.78) | 61.61 (5.87) | 58.51 (16.90)
Sympathetic Cardiac Tone - Low Frequency/High Frequency Spectral Power Ratio [Mean (Standard Deviation); unit: ratio: LF (watts/HZ) / HF (watts/Hz)] — Low frequency to high frequency spectral power was assessed via heart rate variability (HRV) power spectral analysis. This index was reported in normalized units. The ECG signal was acquired via PowerLab 16/35 psychophysiological data acquisition system with a sampling rate of 1000 Hz. Hardware setup included an ECG100C amplifier with a 35Hz LPN filter and a .5Hz HP filter. LF spectral power ranged from 0.04-0.15 Hz. HF spectral power ranged from 0.15-0.45 Hz. The ratio is designed to assess degree of sympathetic innervation to the heart.
  ratio: LF (watts/HZ) / HF (watts/Hz) | 1.02 (1.55) | .99 (.84) | .72 (.53) | .91 (1.18)

OUTCOME MEASURES:

1. Primary Outcome: Rosenberg Self-Esteem Scale (RSE).
Description: The Rosenberg Self-Esteem Scale is designed to assess global feelings of self-worth. The RSE includes 10 items (e.g. "I feel that I'm a person of worth'') rated on a four-point scale (1 = strongly disagree, 4 = strongly agree). A total score represents the sum of individual item responses. Scores range from 10 to 40 and higher scores indicate higher levels of self-esteem.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: Mean scores and standard deviations were reported as a function of group and time. Single mean imputation was used to impute all missing scores to reflect a sample size of n=60 per condition (N=180 total) based on participants admitted at the beginning of the trial. The outcome analyses were based on imputed values and therefore, overall number of participants analyzed equals 60 per condition in the outcome analyses.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 22.71 (4.71) | 22.50 (4.81) | 22.62 (4.07)

2. Primary Outcome: Rosenberg Self-Esteem Scale (RSE).
Description: as for outcome 1
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 23.55 (4.30) | 25.45 (4.50) | 25.08 (4.57)

3. Primary Outcome: Rosenberg Self-Esteem Scale (RSE).
Description: as for outcome 1
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 24.55 (4.74) | 25.55 (4.09) | 26.60 (4.48)

4. Primary Outcome: Eating Disorder Examination Questionnaire (EDE-Q).
Description: The 28-item Eating Disorder Examination Questionnaire global score was used to measure eating disorder symptomatology. Participants report symptomatology over the past 28 days on a 7-point Likert scale from 0 (no days) to 6 (everyday). The EDE-Q contains 4 subscales: Restraint, Weight Concern, Eating Concern, and Shape Concern. Subscale scores are calculated by finding the averages of the subscale items. A global score is also calculated by averaging the subscale scores. Scores range from 0 to 6; higher scores indicate higher levels of eating disorder pathology.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 4.25 (.8) | 3.93 (1.15) | 3.96 (1.02)

5. Primary Outcome: Eating Disorder Examination Questionnaire (EDE-Q).
Description: as for outcome 4
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 4.17 (.64) | 2.93 (1.20) | 3.07 (1.23)

6. Primary Outcome: Eating Disorder Examination Questionnaire (EDE-Q).
Description: as for outcome 4
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 3.74 (.89) | 2.73 (1.20) | 2.78 (1.14)

7. Primary Outcome: Body Shape Questionnaire (BSQ).
Description: The Body Shape Questionnaire (BSQ) was used to measure body dissatisfaction in the present trial. The BSQ is a 34-item scale. Items are measured on a 6-point Likert scale designed to assess the frequency of negative body-related thoughts (1= never, 6 = always). Individual items are summed to compute an overall score. Scores on this scale range from 34 to 204. Higher scores indicate higher frequency of negative body-related thoughts and higher levels of body dissatisfaction.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 139.42 (23.92) | 134.37 (30.15) | 134.73 (28.32)

8. Primary Outcome: Body Shape Questionnaire (BSQ).
Description: as for outcome 7
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 137.65 (20.91) | 110.96 (33.39) | 114.50 (30.96)

9. Primary Outcome: Body Shape Questionnaire (BSQ).
Description: as for outcome 7
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 129.51 (23.74) | 105.19 (32.23) | 105.29 (28.28)

10. Primary Outcome: Social Comparison Rating Scale (SCRS).
Description: The Social Comparison Rating Scale (SCRS) is an 11-item scale used to assess perception of social rank and social comparison tendencies in the present trial. The scale consists of a series of bipolar adjectives (e.g., inferior/superior) separated by the numbers 1 through 10. For each adjective pair, participants are asked to rank themselves in comparison to others. A score around 60 indicates a person, on average, sees themselves approximately equal to others. Higher scores indicate higher levels of favorable social comparison and higher perceived social rank.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 45.59 (17.10) | 43.83 (13.18) | 43.00 (13.80)

11. Primary Outcome: Social Comparison Rating Scale (SCRS).
Description: as for outcome 10
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 51.02 (16.34) | 51.09 (11.68) | 47.35 (14.82)

12. Primary Outcome: Social Comparison Rating Scale (SCRS).
Description: as for outcome 10
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 46.28 (17.39) | 53.39 (10.93) | 53.18 (15.88)

13. Primary Outcome: Self-Objectification Questionnaire (SOQ)
Description: The Self-Objectification Questionnaire (SOQ) is a 10-item self-report inventory designed to assess the relative importance of body competence versus body appearance in sense of self. Participants rank appearance- versus competence-based attributes from 0 to 9 with higher scores representing higher importance. An overall trait self-objectification score is computed by summing competence and appearance ratings and subtracting the sum of competence ratings from the sum of appearance ratings. Resulting scores range from -25 to 25. Higher scores denote higher levels of trait self-objectification.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 10.13 (9.75) | 7.71 (13.11) | 6.32 (12.46)

14. Primary Outcome: Self-Objectification Questionnaire (SOQ)
Description: as for outcome 13
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 10.40 (9.08) | 6.70 (11.39) | 2.35 (13.65)

15. Primary Outcome: Self-Objectification Questionnaire (SOQ)
Description: as for outcome 13
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 9.80 (8.34) | 2.81 (12.39) | 1.78 (12.61)

16. Primary Outcome: Ideal Body Stereotype Scale - Revised.
Description: The Ideal Body Stereotype Scale - Revised was used to assess the extent to which participants internalized the cultural feminine thin-ideal. The IBSS-R is a self-report inventory which asks participants to report their level of agreement with 6 statements which indicate what attractive women look like on a 5-point scale ranging from strongly disagree (1) to strongly agree (5). Responses are averaged to compute a total score. Scores ranges from 1 to 5; higher scores indicate higher levels of thin-ideal internalization.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 3.81 (0.5) | 3.82 (.45) | 3.76 (.5)

17. Primary Outcome: Ideal Body Stereotype Scale - Revised.
Description: as for outcome 16
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 3.76 (0.47) | 3.39 (.69) | 3.60 (.54)

18. Primary Outcome: Ideal Body Stereotype Scale - Revised.
Description: as for outcome 16
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 3.76 (.52) | 3.34 (.59) | 3.46 (.40)

19. Primary Outcome: State Trait Anxiety Inventory - Form Y.
Description: The State Trait Anxiety Inventory- Form Y (STAI) is a 20-item self-report measure used to assess level of trait anxiety in the present study. Each item consists of a statement which assesses feelings of anxiety or relaxation on a 4-point scale ranging from 1 (not at all) to 4 (very much so). Responses to individual items are summed to create an overall score. Scores range from 20 to 80. Higher scores indicate higher levels of anxiety.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 58.87 (8.42) | 58.02 (7.84) | 58.70 (7.90)

20. Primary Outcome: State Trait Anxiety Inventory - Form Y.
Description: as for outcome 19
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 57.15 (7.39) | 53.05 (8.22) | 54.63 (9.31)

21. Primary Outcome: State Trait Anxiety Inventory - Form Y.
Description: as for outcome 19
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 55.63 (9.45) | 51.63 (7.00) | 52.58 (9.71)

22. Primary Outcome: Positive and Negative Affect Scale - Positive Affect
Description: The Positive and Negative Affect Schedule is a 20-item self-report questionnaire that used to measure positive and negative affect. Items are rated on a 5-point scale ranging from 1 (very slightly) to 5 (extremely) which measures the extent to which the client has experienced that affect over the past week. The 10 positive and 10 negative items are summed separately to create a positive affect score and a negative affect score respectively. Each score ranges between 0 and 50 with higher scores indicating higher positive or negative affect.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 26.35 (5.76) | 25.53 (7.10) | 25.24 (6.46)

23. Primary Outcome: Positive and Negative Affect Scale - Positive Affect
Description: as for outcome 22
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 25.54 (6.36) | 28.57 (5.64) | 27.82 (6.69)

24. Primary Outcome: Positive and Negative Affect Scale - Positive Affect
Description: as for outcome 22
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 26.60 (6.44) | 27.84 (5.85) | 27.98 (5.26)

25. Primary Outcome: Mean R Wave Amplitude
Description: Mean R wave amplitude was determined via a 3-lead ECG and was measured in millivolts (mV). The ECG signal was acquired via PowerLab 16/35 psychophysiological data acquisition system with a sampling rate of 1000 Hz. Hardware setup included an ECG100C amplifier with a 35Hz LPN filter and a .5Hz HP filter. ECG data were analyzed via PowerLab LabChart 8 software. A total of 5 minutes and 30 seconds of ECG data were collected to allow for artifact trimming. Artifacts were flagged by experimenters during data collection. Mean R wave amplitude represents ventricular depolarization. Higher magnitudes indicated increased polarity associated with an increased force of ventricular contraction.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
millivolts (mV) | 1.27 (.36) | 1.19 (.31) | 1.27 (.36)

26. Primary Outcome: Mean R Wave Amplitude
Description: Mean R wave amplitude was determined via a 3-lead ECG and was measured in millivolts (mV). The ECG signal was acquired via PowerLab 16/35 psychophysiological data acquisition system with a sampling rate of 1000 Hz. Hardware setup included an ECG100C amplifier with a 35Hz LPN filter and a .5Hz HP filter. ECG data were analyzed via PowerLab LabChart 8 software. A total of 5 minutes and 30 seconds of ECG data were collected to allow for artifact trimming. Artifacts were flagged by experimenters during data collection. Mean R wave amplitude represents ventricular depolarization and is measured in millivolts. Higher magnitudes indicated increased polarity associated with an increased force of ventricular contraction.
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
millivolts (mV) | 1.32 (.32) | 1.19 (.24) | 1.27 (.36)

27. Primary Outcome: Mean R Wave Amplitude
Description: as for outcome 26
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: millivolts (mV)
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
millivolts (mV) | 1.26 (.31) | 1.14 (.26) | 1.12 (.26)

28. Primary Outcome: QT Interval Length
Description: QTc prolongation was measured in msec and was assessed via 3-lead ECG. The ECG signal was acquired via PowerLab 16/35 psychophysiological data acquisition system with a sampling rate of 1000 Hz. Hardware setup included an ECG100C amplifier with a 35Hz LPN filter and a .5Hz HP filter. ECG data were analyzed via PowerLab LabChart 8 software. For detection, typical QRS width was set at 80ms and R waves were at least 300ms apart. QTc was corrected with Bazett's formula. QT interval length represents the length of ventricular depolarization and repolarization and is measured in msec.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
msec | .38 (.02) | .38 (.02) | .38 (.02)

29. Primary Outcome: QT Interval Length
Description: as for outcome 28
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
msec | .38 (.02) | .39 (.01) | .39 (.01)

30. Primary Outcome: QT Interval Length
Description: Mean scores and standard deviations were reported as a function of group and time. Single mean imputation was used to impute all missing scores to reflect a sample size of n=60 per condition (N=180 total) based on participants admitted at the beginning of the trial. The outcome analyses were based on imputed values and therefore, overall number of participants analyzed equals 60 per condition in the outcome analyses.
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
msec | .38 (.02) | .38 (.01) | .38 (.01)

31. Primary Outcome: Vagal Cardiac Tone - High Frequency Spectral Power
Description: High frequency spectral power was assessed via heart rate variability (HRV) power spectral analysis of 3-lead ECG data and was reported in normalized units. The ECG signal was acquired via PowerLab 16/35 psychophysiological data acquisition system with a sampling rate of 1000 Hz. Hardware setup included an ECG100C amplifier with a 35Hz LPN filter and a .5Hz HP filter. ECG data were analyzed via PowerLab LabChart 8 software. Maximum frequency was set at 0.5 Hz with number of frequencies at 500. LF spectral power ranged from 0.04-0.15 Hz. HF spectral power ranged from 0.15-0.45 Hz. Increased high frequency spectral power represents increased vagal input to the heart.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Normalized units: HF (watts/Hz)
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
Normalized units: HF (watts/Hz) | 60.08 (19.56) | 57.26 (19.78) | 61.61 (5.87)

32. Primary Outcome: Vagal Cardiac Tone - High Frequency Spectral Power
Description: as for outcome 31
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Normalized units: HF (watts/Hz)
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
Normalized units: HF (watts/Hz) | 60.15 (21.20) | 60.04 (23.46) | 60.58 (17.52)

33. Primary Outcome: Vagal Cardiac Tone - High Frequency Spectral Power
Description: as for outcome 31
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: Normalized units: HF (watts/Hz)
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
Normalized units: HF (watts/Hz) | 51.65 (20.56) | 56.60 (22.83) | 58.81 (19.68)

34. Primary Outcome: Sympathetic Cardiac Tone - Low Frequency High Frequency Spectral Power Ratio
Description: Low frequency to high frequency spectral power was assessed via heart rate variability (HRV) power spectral analysis of 3-lead ECG. This index was reported in normalized units. The ECG signal was acquired via PowerLab 16/35 psychophysiological data acquisition system with a sampling rate of 1000 Hz. Hardware setup included an ECG100C amplifier with a 35Hz LPN filter and a .5Hz HP filter. Maximum frequency was set at 0.5 Hz with number of frequencies at 500. LF spectral power ranged from 0.04-0.15 Hz. HF spectral power ranged from 0.15-0.45 Hz. The ratio is designed to assess degree of sympathetic innervation to the heart.
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio: LF (watts/HZ) / HF (watts/Hz)
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
ratio: LF (watts/HZ) / HF (watts/Hz) | 1.02 (1.55) | .99 (.84) | .72 (.53)

35. Primary Outcome: Sympathetic Cardiac Tone - Low Frequency High Frequency Spectral Power Ratio
Description: as for outcome 34
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio: LF (watts/HZ) / HF (watts/Hz)
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
ratio: LF (watts/HZ) / HF (watts/Hz) | 1.45 (3.51) | 1.05 (1.17) | .85 (1.02)

36. Primary Outcome: Sympathetic Cardiac Tone - Low Frequency High Frequency Spectral Power Ratio
Description: as for outcome 34
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: ratio: LF (watts/HZ) / HF (watts/Hz)
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
ratio: LF (watts/HZ) / HF (watts/Hz) | 1.54 (1.99) | 1.86 (4.64) | 1.32 (2.84)

37. Primary Outcome: Positive and Negative Affect Scale - Negative Affect
Description: as for outcome 22
Time Frame: Baseline assessments occurred after screening and prior to the delivery of any interventions.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 30.15 (7.46) | 29.00 (6.88) | 29.64 (6.60)

38. Primary Outcome: Positive and Negative Affect Scale - Negative Affect
Description: as for outcome 22
Time Frame: Postintervention assessments were conducted approximately 4 weeks following the baseline assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 29.63 (6.67) | 25.61 (6.99) | 25.59 (6.89)

39. Primary Outcome: Positive and Negative Affect Scale - Negative Affect
Description: as for outcome 22
Time Frame: Follow-up assessments began approximately 8 weeks after the postintervention assessment.
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
Number analyzed (Participants) | 60 | 60 | 60
units on a scale | 28.50 (7.96) | 24.24 (6.24) | 25.00 (5.82)

ADVERSE EVENTS:
Time Frame: Information regarding adverse events were reported at baseline, postintervention (approximately 4 weeks after treatment initiation) and 2-month follow-up (approximately 8 weeks after treatment conclusion).
Arm/Group | Educational Brochure | Body Project Traditional | Body Project Expanded
All-Cause Mortality (participants affected / at risk) | 0/60 | 0/60 | 0/60
Serious Adverse Events (participants affected / at risk) | 1/60 | 0/60 | 2/60
Other Adverse Events (participants affected / at risk) | 0/60 | 0/60 | 0/60
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Educational Brochure (N=60) | Body Project Traditional (N=60) | Body Project Expanded (N=60)
Hospitalization (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0) — Hospitalization
Suicidal Ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03796091/Prot_000.pdf
  • Statistical Analysis Plan (2018-05-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03796091/SAP_001.pdf
  • Informed Consent Form (2018-12-08): https://cdn.clinicaltrials.gov/large-docs/91/NCT03796091/ICF_002.pdf